CLINICAL TRIAL: NCT02251535
Title: Retrospective Non-randomized In-vivo Comparison of Different Levels of Femoral Rollback in the ATTUNE Total Knee Arthroplasiy System on the Basis of Fluoroscopic and Marker-based Motion Capture Evaluation.
Brief Title: In-vivo Comparison of Different Levels of Femoral Rollback in a Primary Total Knee Arthroplasty
Acronym: DePuyAttune
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Carsten Perka (Other)
Collaborators: Julius Wolff Institute (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Carsten Perka, Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DePuy ECO257107
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Gonarthrosis
Keywords: kinematic analysis; femoral rollback; mobile bearing; cruciate retaining Primary Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- test group 1 (Experimental): Retrospective test group 1 (n=10, ATTUNE® Knee System, rotating platform, cruciate retaining) with intraoperative high level rollback
  Interventions: Device: ATTUNE® Knee System
- test group 2 (Experimental): Retrospective test group 2 (n=10, ATTUNE® Knee System, rotating platform, cruciate retaining)with intraoperative low level rollback
  Interventions: Device: ATTUNE® Knee System
- control group (Experimental): Control group (n=10, PFC® SIGMA® Knee System, rotatinq platform, cruciate retaininq)
  Interventions: Device: PFC® SIGMA® Knee System

INTERVENTIONS:
Device: ATTUNE® Knee System
  Arms: test group 1; test group 2
Device: PFC® SIGMA® Knee System
  Arms: control group

SUMMARY:
Retrospective non-randomized in-vivo comparison of different levels of femoral rollback in the ATTUNE total knee arthroplasiy system (rotating platform CR high level roll back vs. rotating platform CR low level roll back) on the basis of fluoroscopic and marker-based motion capture evaluation. How do different levels of intra-operatively observed femoral rollback correlate to postoperative kinematics under weight bearing conditions? Does the modified design of the Attune Knee System influence the extent of the femoral rollback compared to the PFC Sigma Knee System? Does the femoral rollback maintain over a period of 12 months follow up or is it reduced by, for example, remodelling of the posterior cruciate ligament?

DETAILED DESCRIPTION:
Postoperative knee pain is one of the most challenging problems following total knee arthroplasty. Of all the possible complications, the patella-femoral joint is an important cause of postoperative knee pain and prosthetic failure. Nägerl et al. observed that the tibia slides along the femoral surface when the knee is flexed [Nagerlet al., 2009]. Beside the stabilization of the flexion gap, the main task of the posterior cruciate ligament is to initiate the femoral rollback to reduce the patellofemoral pressure. Vice versa, Heyse et al. could show that the patello-femoral pressure rises with the nsuffictency of the posterior cruciate ligament [Heyse et al., 2010]. Pandit et al. measured the physiological rollback in healthy knees and following implantation of currently available TKA. They could show that bonventional TKA are not able to restore the rollback in the natural tibio-femoral joint [Pandit et al., 2005]. Thus it would be important to see if the knee stability in joint replacement reaches the one found in intact or reconstructed knees after surgery. To mimic the femoral rollback a new prosthesis has recently been developed and is about to be introduced to be a new option for total knee arthroplasty. The "Attune Knee System" (DePuy, Warsaw, USA) also has a reduced femoral flange to reduce the patella-femoral contact pressure. The increased rotational stability, the reduced femoral flange and the femoral rollback of the "Attune Knee System" are intended to decrease postoperative knee pain. Different levels of femoral rollback were observed intra-operatively between the Attune and PFC Sigma system. Yoshiya et al. could show the relation between the posterior cruciate ligament with the femoral rollback [Yoshiya et al. 2005]. Therefore, one can hypothesize that different implant designs in combination with the tension of the PCL produce different extents of femoral rollback, ln order to test in-vivo knee kinematics in patients during active movements, we use motion capture, together with combinations of advanced techniques for assessing skeletal kinematics (including sARA [Ehrig et a1.2007], SCoRE [Ehrig et al.2011] & ocsr [Taytor et at. 2005]), a novet non-invasive approach to evaluate dynamic tibio-femoral motion. The combination of these approaches is now able to provide the accuracy and sensitivity required to analyze movement patterns in a rapid, robust and therefore clinically viable manner. ln order to do so, highly advanced equipment is needed which is available in our laboratory in the Julius Wolff lnstitute. Here, we use an infra-red optical motion capture system (10 T20S cameras, Vicon, Oxford, UK; system accuracy \-0.3-0.5 mm), tracked at120Hz, as well as 2 force plates (AMTI 0R6, Watertown, MA, USA) in order to assess the external forces while performing active movements. With this methodology we are then able to measure the kinematics as well as kinetics in the knee joint [Boeth et al., 2013], especially different levels of femoral rollback in patients with ATTUNE implants, during activities of daily living including walking, jogging, stair ascending/descending, rise a chair, sit down. Furthermore lunge can also be performed with single plane fluoroscopy (BV Pulsera, Philips) with a frequency of 30 Hz. During these measurements, the different extents of femoral rollback in deep flexion (at 105'-125') under weight bearing condiiions will be assessed and compared to the Sigma PFC system. The contact point between the femoral component and the polyethylene inlay will be recorded and compared to standardized postoperative radiographs. Clear specification should be given to the subject in order to avoid unnecessary radiation, for this, at least 3 repetitions without radiation should be performed to guarantee a complete subject's understanding of the procedure. The final position of the foot on the sieps is marked to guarantee a standardization of the procedure. The height of the c-arm of the device is adjusted to the specific shank's height of the subject. During the analysis of the fluoroscopic assessment, model-based RSA software (MEDIS, Leiden, The Netherlands) is used to register CAD models of the meiallic implants to the fluoroscopic images, a registration accuracy of 0.6mm and 0.4' has been reported [Moewis elal.2012].

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Both, male and female
2. MinimumAge: 18 Years
3. Osteoarthritis Kellgren Grad lll or lV
4. Mechanical leg axis between 10'valgus and 10' varus
5. Tibial slope between 0' and 10'
6. BMI< 40, participation consent

Exclusion Criteria:

1. Multidirectional instability of the knee
2. connective tissue diseases (Marfan syndrome, Ehlers-Danlos syndrome, scleroderma)
3. Nervous system diseases (Parkinson, multiple sclerosis, Peripheral neuropathy)
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
tibio-femoral anterior-posterior translation | at 12 months post operative
  We intend to collect tibio-femoral anterior-posterior translation during active movement in order to analyse the different extent of femoral rollback (fluoroscopy and gait analysis including lunge activity) at 12 months post operative. Therefore, the femoral rollback will be classified to high level (l) and low level (ll) according to intraoperatively documented findings and postoperative radiographs.

SECONDARY OUTCOMES:
quality of life | at 12 months post operative
  We intend to collect the following secondary objective data pre operatively and '12 months post operative:
  - PKIP
quality of life | at 12 months post operative
  We intend to collect the following secondary objective data pre operatively and '12 months post operative:
  - KOOS
quality of life | at 12 months post operative
  We intend to collect the following secondary objective data pre operatively and '12 months post operative:
  - WOMAC
quality of life | at 12 months post operative
  We intend to collect the following secondary objective data pre operatively and '12 months post operative:
  - SF 36

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine Berlin Center for Musculoskeletal Surgery Department of Orthopaedics, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Center for Musculoskeletal Surgery — http://cmsc.charite.de/
- See also: Julius Wolff Institute for Biomechanics and Musculoskeletal Regeneration — http://jwi.charite.de/en/